CLINICAL TRIAL: NCT03120884
Title: Intracytoplasmic Sperm Injection in Non-male Factor Infertility in Advanced Maternal Age
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: International Peace Maternity and Child Health Hospital (Other)
Responsible Party: Principal Investigator, He-Feng Huang, President, International Peace Maternity and Child Health Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IPMCH2017001
Record Dates: First submitted 2017-04-16; First posted 2017-04-19 (Actual); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Infertility, Female; ART
MeSH Terms: conditions — Infertility, Female | interventions — Sperm Injections, Intracytoplasmic; Fertilization in Vitro

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IVF (Experimental): embryos are cultured using conventional in vitro fertilization.A maximum of 2 embryos will be transferred for each treatment cycle.
  Interventions: Procedure: IVF
- ICSI (Experimental): embryos are fertilized using ICSI.A maximum of 2 embryos will be transferred for each treatment cycle.
  Interventions: Procedure: ICSI

INTERVENTIONS:
Procedure: ICSI — A technique that involves microinjection of spermatozoa into mature oocytes.
  Other Names: Intracytoplasmic Sperm Injection
  Arms: ICSI
Procedure: IVF — A process of fertilisation where an an egg is combined with sperm outside the body, in vitro.
  Other Names: in vitro fertilization
  Arms: IVF

SUMMARY:
This will be a prospective, randomized (1:1 ratio) clinical trial for non-male factor infertility in advanced maternal age with or without intracytoplasmic sperm injection(ICSI). Qualified 1422 patients are randomized into either of two groups: group A will undergo conventional in-vitro fertilization(IVF)(711 cases), Group B will undergo intracytoplasmic sperm injection (ICSI) (711 cases). All participants will receive the same protocol for ovarian stimulation and standardized luteal phase support.

The target population will be patients with non-male factor infertility aged ≥38years with FSH ≤15. Women with other reasons of infertility (eg. anovulation, endometriosis, and premature ovarian failure) are excluded.

The randomization will take place before controlled ovarian stimulation by a computer randomization system. The accumulated live birth rate , pregnancy complications will be followed up by checking medical records and telephone calls.

ELIGIBILITY:
Inclusion Criteria:

* Female patients ages ≥38 years old with FSH ≤15;
* Spouse with normal sperm analysis according to WHO fifth edition criteria(sperm parameter values: total sperm count of at least 39 million, concentration≥15 × 106/ml, total motility ≥40%, progressive motility ≥32%， strict morphology ≥4% normal forms)；
* Female patients who intended to undergo IVF and had signed a written consent form.

Exclusion Criteria:

* More than three previous IVF cycles (including both failed cycles and cycles that ended in live births)
* Female patients with Ovulation dysfunction related disease, such as endometriosis, polycystic ovarian syndrome(tubal factors are not included); undiagnosed infertility; Female patients who have previously been diagnosed with a uterine abnormality such as a malformed uterus(uterus unicornis, septate uterus, duplex uterus or uterus bicomis), adenomyosis, submucous myoma or intrauterine adhesion;
* Spouse who have experienced recurrent spontaneous abortions (including biochemical pregnancy abortion), defined as three or more previous pregnancy losses;
* Patients or their partners with an abnormal chromosome karyotype not including chromosome polymorphisms, which mainly refer to the variants in the chromosomal heterochromatin region
* the use of donor oocytes or sperm;
* the use of frozen oocytes or sperm;
* Femal patients with medical conditions that contraindicate assisted reproductive technology and/or pregnancy, such as poorly controlled type 1 or type 2 diabetes mellitus; undiagnosed liver disease or dysfunction(based on serum liver enzyme test results); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus or cerebrovascular accident; uncontrolled hypertension or known symptomatic heart disease; history of (or suspected) cervical carcinoma, endometrial carcinoma or breast carcinoma; and undiagnosed vaginal bleeding;
* Spouse with medical conditions that contraindicate assisted reproductive technology and/or pregnancy, such as poorly controlled type 1 or type 2 diabetes mellitus; undiagnosed liver disease or dysfunction(based on serum liver enzyme test results); renal disease or abnormal serum renal function; significant anemia; history of deep venous thrombosis, pulmonary embolus or cerebrovascular accident; uncontrolled hypertension or known symptomatic heart disease;
* Female patients or their partners who are unable to comply with the study Procedures;
* Female patients who had previously been randomized to either of the two study groups in this trial.

Ages: 38 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1422 (Estimated)
Dates: Start 2017-09-01 (Estimated); Primary Completion 2018-09-01 (Estimated); Study Completion 2019-09-01 (Estimated)

PRIMARY OUTCOMES:
accumulated live birth rate | 42 weeks
  This will be based on the outcome of either the ICSI or the outcome of the IVF as will all other secondary outcomes

SECONDARY OUTCOMES:
Fertilization rate | 1 day after fertilization
  Fertilization rate was defined as the percentage of fetal heart beat among total retrieved oocytes
Embryo quality | 3day after fertilization
  Embryo quality was evaluated by microscopy.
clinical pregnancy rate | 35 days after embryo transfer
  Clinical pregnancy was defined as an observation of gestational sac via ultrasonography.
implantation rate | 11-12 weeks after embryo transfer
  Implantation rate was defined as the percentage of fetal heart beat among total transferred embryos at 12 weeks' gestational age.
biochemical pregnancy rate | 2 weeks after embryo transfer
  Biochemical pregnancy was defined as numbers of women with an elevated serum β-hCG level of more than 10 mIU/ml.
pregnancy loss rate | 28 gestational weeks in maximum
  Pregnancy loss is defined as any reason that resulted in failure of an embryo to develop, embryonic or fetal death, or spontaneous expulsion of a pregnancy.
ectopic pregnancy rate | 12 gestational weeks in maximum
  Ectopic pregnancy is defined as an embryo implanted outside the uterine.

CONTACTS AND LOCATIONS:
Overall Officials: He-Feng Huang, MD, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (1):
- International Peace Maternity & Child Health Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
undecided